CLINICAL TRIAL: NCT05570656
Title: Modeling Spinal Mobility in Ankylosing Spondylitis (AS) : Towards New Telekinetic Biomarkers
Brief Title: Modeling Spinal Mobility in Ankylosing Spondylitis: Towards New Telekinetic Biomarkers
Acronym: TELESPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL21_0601
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2022-12

CONDITIONS: Ankylosing Spondylitis
Keywords: rheumatology; Rehabilitation; Bioinformatics; Spondylitis; Motion sensor; XSENS-Awinda
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AS patients (Active Comparator): Evaluation of kinematic parameters by wearing X-Sens sensors in different movements (flexion and extension of the spine, tying shoelaces, picking up an object on the ground, walking, etc.)
  Interventions: Device: XSENS-Awinda
- healthy volunteers (Active Comparator): Evaluation of kinematic parameters by wearing X-Sens sensors in different movements (flexion and extension of the spine, tying shoelaces, picking up an object on the ground, walking, etc.)
  Interventions: Device: XSENS-Awinda

INTERVENTIONS:
Device: XSENS-Awinda — The participant wears inertial sensors X-Sens that measure the kinematic data and the amplitude of joint movements during different movements (flexion and extension of the spine, walking, picking up an object on the ground, tying their shoelaces, getting up from a chair... ) Each movement will be repeated 3 times.
  Participants will also have self-questionnaires to complete (BASDAI and BASFI).
  The exams are carried out on one day.

SUMMARY:
Ankylosing spondylitis (AS) is a chronic inflammatory rheumatic disease that mainly affects the spine and pelvis in its axial form. It is responsible for chronic inflammatory pain and sometimes ankylosis with significant functional retention.

Clinicians need markers capable of precisely measuring the restriction of range of motion in these patients, reflections of the activity and/or sequelae of the disease.

The Inverstigators validated movement markers in the AS by a device including inertial sensors (XSENS) and computer modeling. The accuracy and repeatability of the XSENS-Awinda system compared to the reference measurement system have been demonstrated. The XSENS-Awinda device offers new real-time evaluation possibilities for quantitative gait analysis. This opens the way to new diagnostic tools, prognostics and therapeutic perspectives for the clinician.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic inflammatory rheumatic disease that mainly affects the spine and pelvis in its axial form. It is responsible for chronic inflammatory pain and sometimes ankylosis with significant functional retention. Today, these patients benefit from treatments by biotherapy but the functional monitoring of the therapeutic response is based on the clinical examination, questionnaires, and the measurement of CRP (C reactive Protein).

Clinicians need markers capable of precisely measuring the restriction of range of motion in these patients, reflections of the activity and/or sequelae of the disease. The prevention and/or the restoration of these movement limitations, responsible for gait/attitude/balance disorders, are also among the therapeutic objectives of AS.

In the AS, the synergy between the trunk and the lower limbs is altered with a restriction of the movements of the trunk in the three planes of space. The study of the kinematic variability seems to show a loss of complexity. In addition, MRI morphological examinations are insufficient to assess stiffness and functional disability related to AS.

The investigators validated movement markers in the AS by a device including inertial sensors (XSENS) and computer modeling. The accuracy and repeatability of the XSENS-Awinda system compared to the reference measurement system have been demonstrated. The XSENS-Awinda device offers new real-time evaluation possibilities for quantitative gait analysis. This opens the way to new diagnostic tools, prognostics and therapeutic perspectives for the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* BMI between 18.5 and 30
* Written informed consent
* Same gender and age within +/- 3 years compared to an unmatched AS patient

Inclusion criteria specific to the AS group:

* Age 18-65
* BMI between 18.5 and 30
* Written informed consent
* AS meeting the ASAS (Assessment of Spondylo Arthritis International Society) criteria, i.e. with spinal pain ≥ 3 months old, with an age of diagnosis < 45 years, with:

  * Sacroiliitis on imaging AND ≥ 1 sign of spondylarthritis. OR
  * HLA-B27 (human leukocyte antigen-B27) positive AND ≥ 2 other signs of spondylarthritis

Exclusion Criteria:

* Traumatic, tumoral or infectious low back pain
* History of spinal fracture
* History of lumbar, pelvis, hips, ankles, and/or knees surgery
* Severe scoliosis defined by a Cobb angle > 50°
* Severe impairment of uncorrected visual acuity
* Concomitant pathology responsible for ataxia
* Lumbar arthrodesis of two or more stages
* Pregnant or breastfeeding women
* Patient unable to give consent: patient under guardianship or curators, mentally retarded, dementia, language barrier
* Patient not affiliated to a social security plan
* Patient under legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Variation in spinal angle measurement between APS patients and healthy volunteers | 1 day
  Assess the diagnostic performance of angular measurement in the sagittal plane during flexion and extension of the spine in the diagnosis of AS. spinal angle measurement (in degrees) for both APS patients and healthy volunteers will be compared using a Student's test or Wilcoxon Mann Whitney test depending on the distribution. The diagnostic performances of the different kinematic parameters will be estimated in percentage (%) with their 95% confidence interval.

SECONDARY OUTCOMES:
Percentage of AS activity by BASDAI score | 1 day
  The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) is a questionnaire to calculate the activity index of ankylosing spondylitis.
  Rate the intensity of 5 symptoms during the past week, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence at the highest degree.
  This score is an aid in monitoring ankylosing spondylitis.
Percentage of functional impact of the AS by BASFI score | 1 day
  The BASFI (Bath ankylosing spondylitis functional index) reflects functional impact, that is to say the inability to perform actions of daily living. It contains 10 questions on activities of daily living, which are scored with a rating scale from 0 (no functional impairments) to 10 (maximal impairment) [38] (Box 5.2). The sum score ranges from 0 to 10, with higher values indicating worse functioning.
Percentage of functional impact of the AS by BASMI score | 1 day
  The BASMI (Bath Ankylosing Spondylitis Metrology Index) was established to assess the mobility of the spine and hips.
  It measures :
  * the ear/wall distance
  * head rotation
  * flexion of the trunk
  * trunk flexion to the side
  * the distance between the internal malleolus (at the ankles) during the maximum spread of the legs
  A conversion table allows investigators to give a rating from 0 to 10 for each measurement. The average of the 5 ratings gives the BASMI. It varies from 0 to 10 and the higher the rating, the more limited the movements.
Variation of kinematic parameters of movement between BASFI and sensors | 1 day
  Describe the kinematic parameters of the movements evaluated in the BASFI score through the X Sens sensors.
  Clinical parameters are :
  10 questions on activities of daily living, which are scored with a rating scale from 0 (no functional impairments) to 10 (maximal impairment)
  Kinematic parameters measured with the X sens sensors are :
  * Maximum bending, flexion and rotation angle (degrees)
  * Time up and Go (TUG) ( seconds)
  To establish the correlation between the clinical parameters and the kinematic parameters the investigators will use Spearman or Pearson correlation tests.
percentage of diagnosis concordant between the kinematic parameters of the spine and the diagnosis of AS | 1 day
  Evaluate the diagnostic performance of other kinematic parameters of the spine in the diagnosis of AS.
percentage of diagnosis concordant between the kinematic parameters of the lower limb joints and the diagnosis of AS | 1 day
  Evaluate the diagnostic performance of other kinematic parameters of lower limb joints in the diagnosis of AS.
percentage of correlation between clinical and kinematic parameters | 1 day
  establishing the correlation between clinical parameters and kinematic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Christian JORGENSEN, PU-PH, Principal Investigator — UF of Montpellier
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raychaudhuri SP, Deodhar A. The classification and diagnostic criteria of ankylosing spondylitis. J Autoimmun. 2014 Feb-Mar;48-49:128-33. doi: 10.1016/j.jaut.2014.01.015. Epub 2014 Feb 16. PMID 24534717
- [Background] Dougados M, Sepriano A, Molto A, van Lunteren M, Ramiro S, de Hooge M, van den Berg R, Navarro Compan V, Demattei C, Landewe R, van der Heijde D. Sacroiliac radiographic progression in recent onset axial spondyloarthritis: the 5-year data of the DESIR cohort. Ann Rheum Dis. 2017 Nov;76(11):1823-1828. doi: 10.1136/annrheumdis-2017-211596. Epub 2017 Jul 6. PMID 28684556
- [Background] Wang R, Ward MM. Epidemiology of axial spondyloarthritis: an update. Curr Opin Rheumatol. 2018 Mar;30(2):137-143. doi: 10.1097/BOR.0000000000000475. PMID 29227352
- [Background] Costantino F, Talpin A, Said-Nahal R, Goldberg M, Henny J, Chiocchia G, Garchon HJ, Zins M, Breban M. Prevalence of spondyloarthritis in reference to HLA-B27 in the French population: results of the GAZEL cohort. Ann Rheum Dis. 2015 Apr;74(4):689-93. doi: 10.1136/annrheumdis-2013-204436. Epub 2013 Dec 18. PMID 24351517
- [Background] van der Heijde D, Ramiro S, Landewe R, Baraliakos X, Van den Bosch F, Sepriano A, Regel A, Ciurea A, Dagfinrud H, Dougados M, van Gaalen F, Geher P, van der Horst-Bruinsma I, Inman RD, Jongkees M, Kiltz U, Kvien TK, Machado PM, Marzo-Ortega H, Molto A, Navarro-Compan V, Ozgocmen S, Pimentel-Santos FM, Reveille J, Rudwaleit M, Sieper J, Sampaio-Barros P, Wiek D, Braun J. 2016 update of the ASAS-EULAR management recommendations for axial spondyloarthritis. Ann Rheum Dis. 2017 Jun;76(6):978-991. doi: 10.1136/annrheumdis-2016-210770. Epub 2017 Jan 13. PMID 28087505
- [Background] Dagfinrud H, Kvien TK, Hagen KB. Physiotherapy interventions for ankylosing spondylitis. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD002822. doi: 10.1002/14651858.CD002822.pub3. PMID 18254008
- [Background] Zochling J. Measures of symptoms and disease status in ankylosing spondylitis: Ankylosing Spondylitis Disease Activity Score (ASDAS), Ankylosing Spondylitis Quality of Life Scale (ASQoL), Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI), Bath Ankylosing Spondylitis Global Score (BAS-G), Bath Ankylosing Spondylitis Metrology Index (BASMI), Dougados Functional Index (DFI), and Health Assessment Questionnaire for the Spondylarthropathies (HAQ-S). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S47-58. doi: 10.1002/acr.20575. No abstract available. PMID 22588768
- [Background] Soulard J, Vaillant J, Agier CT, Vuillerme N. Gait characteristics in patients with ankylosing spondylitis: a systematic review. Clin Exp Rheumatol. 2021 Jan-Feb;39(1):173-186. doi: 10.55563/clinexprheumatol/le3bmj. Epub 2020 Oct 5. PMID 33025884
- [Background] Sawacha Z, Carraro E, Del Din S, Guiotto A, Bonaldo L, Punzi L, Cobelli C, Masiero S. Biomechanical assessment of balance and posture in subjects with ankylosing spondylitis. J Neuroeng Rehabil. 2012 Aug 29;9:63. doi: 10.1186/1743-0003-9-63. PMID 22931459
- [Background] Del Din S, Carraro E, Sawacha Z, Guiotto A, Bonaldo L, Masiero S, Cobelli C. Impaired gait in ankylosing spondylitis. Med Biol Eng Comput. 2011 Jul;49(7):801-9. doi: 10.1007/s11517-010-0731-x. Epub 2011 Jan 13. PMID 21229328
- [Background] Robert-Lachaine X, Mecheri H, Larue C, Plamondon A. Accuracy and repeatability of single-pose calibration of inertial measurement units for whole-body motion analysis. Gait Posture. 2017 May;54:80-86. doi: 10.1016/j.gaitpost.2017.02.029. Epub 2017 Mar 1. PMID 28279850
- [Background] Iosa M, Picerno P, Paolucci S, Morone G. Wearable inertial sensors for human movement analysis. Expert Rev Med Devices. 2016 Jul;13(7):641-59. doi: 10.1080/17434440.2016.1198694. Epub 2016 Jun 17. PMID 27309490